CLINICAL TRIAL: NCT00943501
Title: Liraglutide: A Randomized, Double-blind, Placebo Controlled Trial to Assess Safety/Tolerability, Pharmacokinetics & Pharmacodynamics of Liraglutide in Pediatric (10-17 Years Old) With Type 2 Diabetes
Brief Title: Safety of Liraglutide in Pediatric Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1800; U1111-1111-9256 (Other: WHO); 2010-021057-39 (EudraCT Number)
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- I.a (Experimental)
  Interventions: Drug: liraglutide
- I.b (Placebo Comparator)
  Interventions: Drug: placebo
- II.a (Experimental)
  Interventions: Drug: liraglutide
- II.b (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — Increasing dose for self-injection subcutaneously (under the skin) daily over 5 weeks (0.3 - 1.8 mg)
  Arms: I.a
Drug: placebo — Increasing dose for self-injection subcutaneously (under the skin) daily over 5 weeks (0.3 - 1.8 mg)
  Arms: I.b
Drug: liraglutide — Increasing dose for self-injection subcutaneously (under the skin) daily over 3 to 4 weeks (0.6 - 1.8 mg).
  Arms: II.a
Drug: placebo — Increasing dose for self-injection subcutaneously (under the skin) daily over 3 to 4 weeks (0.6 - 1.8 mg).
  Arms: II.b

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this clinical trial is to investigate the safety, tolerability, pharmacokinetics (the determination of the concentration of the administered medication in blood over time) and pharmacodynamics (the determination of the effect over time and the duration of action) of multiple doses of liraglutide in the pediatric population (children).

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than 85th percentile for age and gender
* Currently being treated with diet and exercise or metformin alone
* HbA1c (glycosylated haemoglobin) between 6.5 and 11.0%

Exclusion Criteria:

* Any clinically significant disease other than type 2 diabetes, as judged by the trial physician
* Previous treatment with any anti-diabetic drug other than metformin (except for prior short term treatment, at the discretion of the trial physician)

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse events | up to 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration vs. time curve | within dosing interval
Pharmacodynamics: Fasting Plasma Glucose (FPG) and insulin | throughout study duration (pre-, during and post-treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (19):
- United States (13):
  - Novo Nordisk Investigational Site, Cypress, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Toledo, Ohio
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
- Novo Nordisk Investigational Site, Brussels, Belgium
- Novo Nordisk Investigational Site, Ljubljana, Slovenia
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Result] Klein DJ, Battelino T, Chatterjee DJ, Jacobsen LV, Hale PM, Arslanian S; NN2211-1800 Study Group. Liraglutide's safety, tolerability, pharmacokinetics, and pharmacodynamics in pediatric type 2 diabetes: a randomized, double-blind, placebo-controlled trial. Diabetes Technol Ther. 2014 Oct;16(10):679-87. doi: 10.1089/dia.2013.0366. Epub 2014 Jul 18. PMID 25036533
- [Result] Petri KC, Jacobsen LV, Klein DJ. Comparable liraglutide pharmacokinetics in pediatric and adult populations with type 2 diabetes: a population pharmacokinetic analysis. Clin Pharmacokinet. 2015 Jun;54(6):663-70. doi: 10.1007/s40262-014-0229-z. PMID 25603819
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com